CLINICAL TRIAL: NCT06714890
Title: A Single-center, Prospective, Randomized Controlled Trial Evaluating Accommodation-related Visual Training Combined with Transcranial Electrical Stimulation Versus Accommodation-related Visual Training Alone for the Treatment of Accommodation Dysfunction
Brief Title: Accommodation-Related Visual Training Combined with Transcranial Electrical Stimulation Versus Visual Training Alone for the Treatment of Accommodation Dysfunction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-tES
Record Dates: First submitted 2024-12-02; First posted 2024-12-04 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia; Esotropia
Keywords: Acute Acquired Concomitant Esotropia; Presbyopia; Accommodation Disorder; Transcranial Electrical Stimulation; Visual Training
MeSH Terms: conditions — Presbyopia; Esotropia | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial Electrical Stimulation Group (Experimental): visual training combined with transcranial electrical stimulation
  Interventions: Device: Transcranial Electrical Stimulation
- Visual Training Group (Active Comparator): visual training
  Interventions: Other: Visual Training

INTERVENTIONS:
Device: Transcranial Electrical Stimulation — Transcranial Electrical Stimulation Combined with Accommodation-related Visual Training
  Arms: Transcranial Electrical Stimulation Group
Other: Visual Training — Accommodation-related Visual Training
  Arms: Visual Training Group

SUMMARY:
This is a single-center, randomized controlled trial to compare the effectiveness of transcranial electrical stimulation combined with visual training with visual training alone for the treatment of accommodation disorder patients.

DETAILED DESCRIPTION:
Accommodation is a dynamic process in which the eyes focus on targets at different distances. When the human eye turns its gaze point from far to near, the lens, ciliary body, and suspensory ligament need to work in coordination to make the object clearly imaged on the retina. Clinically, the occurrence and development of many ophthalmic diseases are related to accommodative dysfunction. This study mainly focuses on two types of accommodative eye diseases, presbyopia and acute acquired concomitant esotropia (AACE).

More than 1 billion adults worldwide are affected by presbyopia, and some studies believe that the occurrence of presbyopia is mainly related to the decline of accommodative function. Accommodative visual training can improve the symptoms of presbyopia, but there are problems such as long treatment course, great impact on daily life, and poor patient compliance. AACE is another eye disease related to accommodative dysfunction. AACE is a relatively rare type of esotropia, but the incidence has shown a significant upward trend in recent years. Scholars believe that its high incidence is mainly related to the increased accommodative load when the eyes are used excessively at close range. Studies have found that AACE at the early stage of onset and at a small angle can reduce the degree of strabismus through visual training related to accommodation, but the recovery of accommodation function and strabismus will have a plateau period, and patients have poor compliance with training. Since the existing treatment for accommodation dysfunction, namely visual training, has problems such as long treatment course, great impact on daily life, and poor compliance, it is necessary to explore more effective alternative treatment methods with lower compliance requirements to better serve the needs of patients.

Electrical stimulation treatment is very safe and is a non-invasive treatment method. By placing electrodes on specific brain areas and applying weak currents to the scalp, the state of brain activity is changed. This method has been widely used in other mental disorders. At present, in the field of ophthalmology, some scholars have used transcranial electrical stimulation to treat patients with amblyopia and convergence insufficiency, and found that electrical stimulation can improve patients' contrast sensitivity, stereoscopic vision and convergence function. The above studies have proved the application prospects of transcranial electrical stimulation in visual diseases, which can be used to treat visual diseases by reshaping the functions related to the visual nerve. Regarding the accommodation function, some scholars have also found that transcranial electrical stimulation can affect the accommodation function of the eye lens by changing the excitability of the visual cortex. In addition, magnetic resonance imaging studies have found brain areas related to accommodation function, including the frontal eye movement area and occipital lobe, which can be used as sites for electrical stimulation. Therefore, for patients with abnormal accommodation function, transcranial electrical stimulation therapy may be a promising treatment method. It can not only reshape the function of accommodation-related nerves, but also has the advantages of short treatment course, low compliance requirements, and no impact on patients' daily life. It can also make up for the disadvantages of visual training.

When exploring the potential effects of electrical stimulation combined with visual training on patients with abnormal accommodation function, functional magnetic resonance imaging (fMRI) technology will play a key role. Accommodation is a cause of many eye diseases, and there is little exploration of the brain area of accommodation function. Existing research on accommodation function focuses on the physiological structural changes of the lens and ciliary muscle. Through fMRI research, we can explore the activity changes and remodeling of the accommodation-related visual pathways in patients with abnormal accommodation function after receiving tDCS in a more in-depth and intuitive way.

Based on scientific research findings, tES combined with visual tasks can reshape the accommodative function, but no studies have fully explored the effectiveness and safety of this method in treating patients with abnormal accommodative function, nor have studies compared the therapeutic effects of visual training and tES combined with visual tasks on patients with abnormal accommodative function. In order to better guide clinical practice, we plan to conduct a randomized controlled study to objectively evaluate and compare the therapeutic effects of visual training and transcranial electrical stimulation combined with visual tasks on patients with abnormal accommodative function, and to conduct in-depth research on the remodeling of brain areas related to accommodation through fMRI technology. It is expected that the research results will provide more treatment options for patients with abnormal accommodative function, and provide important guidance for the clinical selection of appropriate methods to treat patients with abnormal accommodative function.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion criteria for small-angle acute concomitant esotropia: clinical diagnosis of acute aquired concomitant esotropia; strabismus angle ≤ 15PD; age 18 < age < 40; best corrected visual acuity of both eyes ≥ 1.0.
2. Inclusion criteria for presbyopia: clinical diagnosis of presbyopia; best corrected visual acuity of both eyes ≥ 1.0.

Exclusion Criteria:

1. no history of other eye diseases or eye surgeries
2. no history of neuropsychiatric diseases for the individual or relatives
3. no head injuries or surgeries
4. no history of epilepsy or stroke
5. no metal implants in the body
6. no claustrophobia, no metal implants in the body (fracture fixation nails, pacemakers, etc.)
7. pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Amplitude of Accommodation | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  using minus lens method to evaluate amplitude of accommodation
Accommodation Response | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  using binocular cross-cylinder method to evaluate accommodation response
Positive and negative relative accommodation | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  using phoropter examination to evaluate positive and negative relative accommodation
Accommodation Facility | Before treatment, 1 week, 1 month, 3 months, 6 months after treatment
  Using flipper to evaluate the accommodation facility

CONTACTS AND LOCATIONS:
Overall Officials: Wen Wen, MD, PhD, Study Chair — Eye & ENT Hospital of Fudan University, Shanghai, China
Locations (1):
- Eye & ENT Hospital of Fudan University, Shanghai, China, China

IPD SHARING:
Plan to Share IPD: No
We concerns about patient privacy issues and it iss better to protect the publication potential.